CLINICAL TRIAL: NCT00791908
Title: Comparison of Electrodessication, Potassium Titanyl Phosphate (KTP) Laser and Pulsed Dye Laser for Treatment of Cherry Angiomata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Murad Alam, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MA-STU81
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Cherry Angioma
MeSH Terms: interventions — Lasers, Dye; potassium titanylphosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- electrodessication (ED) (Experimental): Treatment over 6 weeks using electrodessication (ED) to remove cherry angiomas. Each participant received treatment with PDL, KTP laser, and electrodesiccation to separate randomly selected areas on the torso, with each area bearing 4 cherry angiomata.
  Interventions: Procedure: Electrodessication
- pulsed dye laser (PDL) (Experimental): Treatment over 6 weeks using pulsed dye laser (PDL) to remove cherry angiomas. Each participant received treatment with PDL, KTP laser, and electrodesiccation to separate randomly selected areas on the torso, with each area bearing 4 cherry angiomata.
  Interventions: Procedure: Pulsed dye laser (PDL)
- potassium titanyl phosphate (KTP) laser (Experimental): Treatment over 6 weeks using potassium titanyl phosphate (KTP) laser to remove cherry angiomas. Each participant received treatment with PDL, KTP laser, and electrodesiccation to separate randomly selected areas on the torso, with each area bearing 4 cherry angiomata.
  Interventions: Procedure: potassium titanyl phosphate (KTP)

INTERVENTIONS:
Procedure: Electrodessication — Treatment applied to a third of the torso at each study visit.
  Arms: electrodessication (ED)
Procedure: Pulsed dye laser (PDL) — Laser treatment applied to a third of the torso at each study visit.
  Arms: pulsed dye laser (PDL)
Procedure: potassium titanyl phosphate (KTP) — Laser treatment applied to a third of the torso at each study visit.
  Arms: potassium titanyl phosphate (KTP) laser

SUMMARY:
The primary objective of this study is to determine whether laser treatments over 6 weeks using the pulsed dye laser system or the potassium titanyl phosphate (KTP) laser are effective in patients with cherry angiomas as observed by a physician provider and the subject.

The investigators hypothesize that the two laser treatments will be an effective tool for treating cherry angiomas. The investigators aim to compare these modalities to electrodessication, as all three modalities are considered the current standard of care. Electrodessication can result in atrophic lesions at the site of the treated cherry angiomas.

In summary, the goal of this project is to compare the non-ablative pulsed dye laser and the AuraTM potassium titanyl phosphate (KTP) laser to each other and to the current standard of care, electrodessication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 95 years.
* Have at least 12 cherry angiomas (4 per each third of the torso) that have been documented.
* The subjects are in medically stable condition.
* The subject has willingness and the ability to understand and provide informed consent for the procedure and is able to communicate with the investigator.
* Must be willing not to employ other treatment options for cherry angiomas during the course of this study.

Exclusion Criteria:

* Under 18 years of age and over 95 years of age
* Pregnancy or lactation.
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects cannot have had previous laser treatment in the last 6 months before enrollment.
* Subjects have a cardiac defibrillator or pacemakers that may interact with the electrodesiccation technique.
* Subjects have no serious medical conditions that would contradict participation in the research.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Collyer J, Boone SL, White LE, Rademaker A, West DP, Anderson K, Kim NA, Smith S, Yoo S, Alam M. Comparison of treatment of cherry angiomata with pulsed-dye laser, potassium titanyl phosphate laser, and electrodesiccation: a randomized controlled trial. Arch Dermatol. 2010 Jan;146(1):33-7. doi: 10.1001/archdermatol.2009.318. PMID 20083690

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes in Color, Texture, and Size of Cherry Angiomata From Baseline to 3 Months After the Second Treatment by Treatment Type as Assessed by Blinded Raters
Description: Each subject received all 3 treatments. Serial standardized photographs evaluated for color,texture and size by 2 blinded dermatologists using ordinal visual analog scales from 0 to 10(color: 0=skin colored, 5=red, 10=purple; texture: 0=flat, 5=mildly elevated, 10=elevated; size: 0=0mm, 10=10 mm).
Time Frame: Baseline and 3 months
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Electrodesiccation (ED); KTP Laser; Pulsed-dye Laser (PDL): Laser treatment applied to a third of the torso at each study visit.
Arm/Group | Electrodesiccation (ED) | KTP Laser | Pulsed-dye Laser (PDL)
Number analyzed (Participants) | 15 | 15 | 15
Units on a scale
  Color of Cherry Angiomata | 5.27 [0 to 10] | 4.99 [0 to 10] | 5.19 [0 to 10]
  Texture of Cherry Angiomata | 4.24 [0 to 10] | 3.42 [0 to 10] | 3.24 [0 to 10]
  Size of Cherry Angiomata | 3.40 [0 to 10] | 3.44 [0 to 10] | 3.31 [0 to 10]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Electrodesiccation (ED) | KTP Laser | Pulsed-dye Laser (PDL)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Absence of a cost analysis; all the participants were white; only one set of parameters (ie, for lasers, pulse duration and fluence; and for electrodesiccation, energy level) was used for treatment with each modality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No